CLINICAL TRIAL: NCT03029104
Title: Collagen Cross-Linking With Ultraviolet-A in Asymmetric Corneas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sufficient clinical results obtained to support study endpoints.
Sponsor: Cxlusa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CXL-005
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Keratoconus; Corneal Diseases; Eye Diseases; Photosensitizing Agents
Keywords: Keratoconus; Forme fruste keratoconus; Post-LASIK ectasia; Pellucid marginal degeneration; Forme fruste pellucid marginal degeneration; Diurnal fluctuation post-radial keratotomy; Terrien's marginal degeneration
MeSH Terms: conditions — Keratoconus; Corneal Diseases; Eye Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Visual acuity will be evaluated by an observer who is masked as to the treatment protocol to which study subjects have been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Group 1 (Active Comparator): Ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) using CXLO Corneal Strengthening Solution and a UVA irradiance of 4 mW/cm2 cycled On/Off at 15 second intervals for 20 minutes.
  Interventions: Combination Product: CXLO Corneal Strengthening Solution and UVA Illumination Device
- Group 2 (Active Comparator): Ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) using CXLO Corneal Strengthening Solution and a UVA irradiance of 6 mW/cm2 cycled On/Off at 15 second intervals for 20 minutes.
  Interventions: Combination Product: CXLO Corneal Strengthening Solution and UVA Illumination Device
- Group 3 (Active Comparator): Ultraviolet-A (UVA)-induced cross-linking of corneal collagen (CXL) using CXLO Corneal Strengthening Solution and a UVA irradiance of 4 mW/cm2 cycled On/Off at 15 second intervals for 30 minutes.
  Interventions: Combination Product: CXLO Corneal Strengthening Solution and UVA Illumination Device

INTERVENTIONS:
Combination Product: CXLO Corneal Strengthening Solution and UVA Illumination Device — CXLO Corneal Strengthening Solution

SUMMARY:
This study will assess changes in visual acuity and corneal symmetry after corneal collagen cross-linking (CXL) of asymmetric corneas.

DETAILED DESCRIPTION:
This study will evaluate the results of Corneal Collagen Crosslinking (CXL) in patients with conditions that include keratoconus, forme fruste keratoconus, post-LASIK ectasia, pellucid marginal degeneration, forme fruste pellucid marginal degeneration, diurnal fluctuation post-radial keratotomy, or Terrien's marginal degeneration. This is an outcomes study, all patients receive treatment.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of at least one of the following conditions:

  1. Keratoconus
  2. Forme fruste keratoconus
  3. Post-LASIK ectasia
  4. Pellucid marginal degeneration
  5. Forme fruste pellucid marginal degeneration
  6. Diurnal fluctuation post-radial keratotomy
  7. Terrien's marginal degeneration

Exclusion Criteria:

1. Corneal thickness < 375 microns measured by ultrasound or Pentacam.
2. Contraindications or hypersensitivities to any study medications or their components.
3. Pregnancy or breastfeeding.
4. Any history of herpes simplex corneal disease in an eye to be treated.
5. Nystagmus or any other condition that would, in the judgement of the investigator, prevent a steady gaze during the treatment.
6. Inability to cooperate with diagnostic tests.
7. Enrollment in another ophthalmic clinical trial.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2228 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2020-12-27 (Actual); Study Completion 2020-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg J Berdy, MD, FACS, Principal Investigator — Ophthalmology Associates, St. Louis, MO
Locations (9):
- United States (9):
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Goodman Eye Center, San Francisco, California
  - Cornea Consultants of Colorado, Littleton, Colorado
  - Woolfson Eye Institute, Atlanta, Georgia
  - Chicago Cornea Consultants, Chicago, Illinois
  - Chicago Cornea Consultants, Ltd., Hoffman Estates, Illinois
  - Ophthalmology Associates, St Louis, Missouri
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Cornea Associates of Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Epstein RJ, Belin MW, Gravemann D, Littner R, Rubinfeld RS. EpiSmart Crosslinking for Keratoconus: A Phase 2 Study. Cornea. 2023 Jul 1;42(7):858-866. doi: 10.1097/ICO.0000000000003136. Epub 2022 Sep 28. PMID 36173242

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 745 | 735 | 748
Completed | 612 | 597 | 623
Not Completed | 133 | 138 | 125

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 745 | 735 | 748 | 2228
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (13.04) | 32.4 (13.11) | 32.6 (12.94) | 32.5 (13.03)
Age, Customized [Number; unit: participants]
  ≤21 years | 175 | 163 | 175 | 513
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 217 | 220 | 658
  Male | 524 | 518 | 528 | 1570
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 142 | 118 | 138 | 398
  Not Hispanic or Latino | 603 | 617 | 609 | 1829
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 3 | 7
  Asian | 32 | 38 | 31 | 101
  Native Hawaiian or Other Pacific Islander | 3 | 7 | 2 | 12
  Black or African American | 92 | 89 | 99 | 280
  White | 582 | 573 | 584 | 1739
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 34 | 26 | 29 | 89
Region of Enrollment [Number; unit: participants]
  United States | 745 | 735 | 748 | 2228
Diagnosis of Keratoconus [Count of Participants; unit: Participants] | 644 | 635 | 643 | 1922

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Corrected Distance Visual Acuity (CDVA)
Description: Changes in CDVA are reported as the value at 6 and 12 months minus the value at baseline
Time Frame: Baseline and 6 and 12 months
Population: Keratoconus subjects completing assessment
Measure: Mean (Standard Error); unit: logMAR
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 542 | 534 | 529
logMAR
  6 months: number analyzed (Participants) | 472 | 461 | 467
  6 months | -0.058 (0.0088) | -0.068 (0.0094) | -0.064 (0.0104)
  12 months: number analyzed (Participants) | 264 | 247 | 273
  12 months | -0.074 (0.0119) | -0.060 (0.0127) | -0.071 (0.0176)

2. Secondary Outcome: Change From Baseline in Uncorrected Distance Visual Acuity (UCVA)
Description: Changes in UCVA are reported as the value at 6 and 12 months minus the value at baseline
Time Frame: Baseline and 6 and 12 months
Population: Keratoconus subjects completing assessment
Measure: Mean (Standard Error); unit: logMAR
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 541 | 533 | 528
logMAR
  6 months: number analyzed (Participants) | 469 | 461 | 468
  6 months | -0.0853 (0.0150) | -0.1099 (0.0150) | -0.0990 (0.0155)
  12 months: number analyzed (Participants) | 263 | 247 | 272
  12 months | -0.0875 (0.0191) | -0.0696 (0.0197) | -0.1243 (0.0212)

3. Secondary Outcome: Change From Baseline in Maximum Keratometry (KMax)
Description: Kmax is the maximum value of corneal curvature in Diopters. Changes in Kmax are reported as the value at 6 and 12 months minus the value at baseline.
Time Frame: Baseline and 6 and 12 months
Population: Keratoconus subjects completing assessment
Measure: Mean (Standard Error); unit: Diopters
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 542 | 533 | 527
Diopters
  6 months: number analyzed (Participants) | 471 | 460 | 465
  6 months | -0.1979 (0.1069) | -0.4033 (0.1228) | -0.3673 (0.1125)
  12 months: number analyzed (Participants) | 263 | 246 | 270
  12 months | -0.2859 (0.1204) | -0.5268 (0.1716) | -0.5256 (0.1707)

ADVERSE EVENTS:
Time Frame: 12 months
Description: A total of 2,228 subjects were randomized and treated in this study (Treated Analysis Set). 1,583 (71%) of these subjects received bilateral, simultaneous treatments. The Safety Analysis Set (SAS) is larger than the Treated Analysis Set because subjects who had an initial unilateral treatment and then had a subsequent procedure, appear in the SAS under two different treatment groups, if the subsequent treatment differs from the initial treatment. This occurred in 19 subjects.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/750 | 0/745 | 0/752
Serious Adverse Events (participants affected / at risk) | 0/750 | 0/745 | 1/752
Other Adverse Events (participants affected / at risk) | 0/750 | 0/745 | 0/752
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=750) | Group 2 (N=745) | Group 3 (N=752)
Diverticulitis (Infections and infestations) | 0 | 0 | 1 — Subject developed diverticulitis 208 days post-procedure; not related; treated and resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT03029104/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT03029104/SAP_001.pdf